CLINICAL TRIAL: NCT01849757
Title: Comparison of Priming Constituents in Patients Undergoing CPB Assisted Cardiac Surgery: HES 130/0.4 or Albumin 5%
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pentaspan is no longer used at our institution. Pentaspan was an arm of the study
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jo-Anne Marcoux, Perfusionist M. Sc., CPC, CCP, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ruh/westerncan/primestudy
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease; Aortic Valve Disease; Mitral Valve Disease
Keywords: Cardiopulmonary bypass; prime; crystalloid; albumin; HES 130/0.4
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease | interventions — Sodium Chloride; normosol R; Ringer's Lactate; Plasmalyte A; Serum Albumin, Human; zidovudine 5'-monophosphate-mannose-albumin conjugate; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Human Albumin (Active Comparator): Human albumin solution used as part of the priming volume for the cardiopulmonary bypass circuit.
  Interventions: Other: Human Albumin
- Voluven or hydroethylstarch HES 130/0.4 (Active Comparator): Hydroethylstarch HES 130/0.4 used as part of the priming volume for the cardiopulmonary bypass circuit.
  Interventions: Other: Voluven
- Crystalloid (Placebo Comparator): Crystalloid will be used to prime the cardiopulmonary bypass circuit
  Interventions: Other: prime crystalloid

INTERVENTIONS:
Other: prime crystalloid — used for priming the CPB circuit
  Other Names: saline 0.9%; Normosol; Ringer's lactate; Plasmalyte
  Arms: Crystalloid
Other: Human Albumin — Used as a constituent for priming the CPB circuit
  Other Names: Albumin 5%; Albumin 25%
  Arms: Human Albumin
Other: Voluven — Used as a constituent for priming the CPB circuit
  Other Names: Hydroethylstarch HES130/0.4
  Arms: Voluven or hydroethylstarch HES 130/0.4

SUMMARY:
The purpose of the study is to determine which priming fluid is the safest for use for priming the heart-lung machine used during cardiopulmonary bypass for patients undergoing cardiac surgery. The fluids to be compared are albumin and voluven. A control group will receive only crystalloid.

DETAILED DESCRIPTION:
Project title:

Comparison of priming constituents in patients undergoing CPB assisted cardiac surgery: 6% HES 130/0.4 or Albumen 5%

Principal investigator:

Jo-Anne Marcoux M. Sc., CPC, CCP

Department:

Clinical Perfusion

Sub-investigators:

Victor Uppal B. Sc., CPC, CCP Taras Mycyk MD, FRCSC,

Research will be conducted at: the cardiac operating rooms of the Royal University Hospital, and affiliated hospitals

Hypothesis It is hypothesized that the use of an artificial colloid (6% hydroxyethyl starch 130/0.4) (HES) as a priming constituent is more disruptive to the coagulation and renal systems compared to the use of human derived albumen.

It is further hypothesized that patients who undergo cardiopulmonary bypass (CPB) with HES 130/0.4 as a priming constituent will demonstrate decreased creatinine clearance and increased post-operative bleeding and transfusion requirements.

Academic validity Permissive hemodilution results when crystalloids and colloids are substituted for blood as priming fluids in the cardiopulmonary bypass circuit. While there are obvious benefits to decreasing autologous blood exposure to the patients undergoing CPB, determining the most physiological substitution has not been conclusively resolved. Historically, available HES had a greater molecular weight then the product currently in use and was associated with detrimental adverse events when compared to saline as fluid replacement therapy (5.3% vs. 2.8%, p < 0.001). (1) When albumin was compared to HES 450/0.7 and HES 200/0.05 for fluid management in adult CPB surgery, (18 trials of 970 patients) HES increased transfusion of red blood cells by 28.4% (p = 0.027), increased the transfusion of fresh-frozen plasma by 30.6% (p = 0.008) and increased the transfusion of platelets by 29.8% (p = 0.027). HES 130/0.4 could not be compared to albumen in this same study because there was insufficient data collected. However, no significant differences were found when comparing transfusion requirements between HES 450/0.7, HES 200/0.05 and HES 130/0.4. (2) Viscoelastic device analysis concluded that the administration of HES 130/0.4 in patients or healthy volunteers resulted in a weaker and smaller clot. (3) Short-time infusions of HES 200/0.5 and HES 130/0.4 after cardiac surgery produced a temporary impairment of fibrin formation and clot strength while human albumin had no effect. (4)

In regards to the association between HES and renal failure, on the one hand use of HES 130/0.4 as a priming fluid used in children undergoing CPB did not result in any negative effects on renal function and was safe to use in the pediatric population. (5) On the other hand, when used for resuscitative measures in 7000 randomly assigned patients admitted to intensive care, though there was no difference in 90 day mortality between the group assigned HES 130/0.4 and the group assigned saline, more patients assigned HES 130/0.4 required renal replacement therapy. (1) When used immediately after CPB in a double-blind clinical trial comparing 4% gelatin, Ringer's solution and HES 130/0.4, it was found that significantly lower mean creatinine levels were found in the HES 130/0.4 group compared to the other two groups. (6)

Our research is directed toward determining conclusively if HES 130/0.4 has a similar risk profile to HES 450/0.7 and HES 200/0.05 when used as a priming constituent for the CPB circuit. Additionally we will determine if an albumin/crystalloid prime is superior to a HES 130/0.4/crystalloid prime. A fully crystalloid prime control group will be included for a controlled comparison.

Research design/Methods

The will be a randomized, control trial. Three groups of subjects will be studied:

1. Control group: Crystalloid prime

   * 2 L crystalloid prime,
   * 2.5 mL/kg Mannitol 20%,
   * 1 ampoule of NaHCO-3 (50 mL),
   * 10,000 iu heparin
2. Voluven (light?):

   * HES 130/0.4 prime 500 mL
   * balance of crystalloid
   * 2.5 mL/kg Mannitol 20%,
   * 1 ampoule of NaHCO-3 (50 mL),
   * 10,000 iu heparin
3. Albumin:

   * Human albumin 500 mL 5%
   * balance of crystalloid
   * 2.5 mL/kg Mannitol 20%,
   * 1 ampoule of NaHCO-3 (50 mL),
   * 10,000 iu heparin

Statistical Analysis We would like to have 7000 subjects included in this research project. Study populations and outcomes for patients undergoing CPB assisted cardiac surgery are extremely varied. An extremely large population size will be necessary to answer the research question proposed as the priming differences in question result in very subtle outcome differences.

All patients will undergo CPB assisted cardiac surgery. Blood samples will be drawn at routine intervals from each subject. Blood will be sampled upon entering the operating room, at the completion of surgery, and at 24 hours post-operatively.

The amount of blood drawn will not be above and beyond the usual tests and analyses related to the care of all affected patients undergoing CPB assisted cardiac surgery.

a)

Inclusion criteria:

* greater than 50 years of age
* will be afflicted with co-morbidities associated with cardiac disease (increased cholesterol, hypertension, smoking, diabetes, previous myocardial infarctions and decreased ejection fraction)

Exclusion criteria:

* emergencies
* renal failure
* dialysis dependent

The cardiac center involved to date is:

RUH Saskatoon The goal is recruitment of all cardiac centers in western Canada.

Primary end-points: are postoperative bleeding and transfusion of autologous units of red blood cells, frozen plasma and platelets.

Secondary end-points: Post-operative renal function parameter creatinine

Data collection will be ongoing. Interim analysis will be completed once half the patients have been recruited with final statistical analysis to be conducted once data capture is complete.

Potential Significance/Justification CPB assisted cardiac surgical outcomes have improved tremendously since the first such procedure was done in 1953. Outcome improvements have always come from small changes that were evidence based. This research project means to determine the safest prime for a procedure, which occurs roughly 2,000,000/year throughout the world. In regards to the cost of the study solutions in question, there is a $4.10 difference between the cost of 500 mL of HES 130/0.4 prime and 500 mL of 5% Albumin with HES 130/0.4 being more expensive.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing cardiopulmonary bypass assisted cardiac surgery

-

Exclusion Criteria:

emergencies and patients in renal failure or dialysis -

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative bleeding and transfusion requirements | 24-48 hours post-operatively
  Postoperative cardiac patients have chest tubes in place which drain any blood oozing from around the pericardial cavity. The chest tubes are attached to a blood collection apparatus which measures the amount of blood loss. Too much post-operative blood loss results in a transfusion requirement of red blood cells, plasma and/or platelets.

SECONDARY OUTCOMES:
renal function, creatinine levels | 24-48 hours post-operatively
  Use of some colloids have been associated with a deterioration of renal function. Data will be collected post-operatively to determine he effect of the different priming fluids on renal function

CONTACTS AND LOCATIONS:
Overall Officials: Jo-Anne E Marcocoux, M. Sc., Principal Investigator — Royal University Hospital Foundation; Jo-Anne E Marcoux, M. Sc., Principal Investigator — RUH
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Myburgh JA, Finfer S, Bellomo R, Billot L, Cass A, Gattas D, Glass P, Lipman J, Liu B, McArthur C, McGuinness S, Rajbhandari D, Taylor CB, Webb SA; CHEST Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Hydroxyethyl starch or saline for fluid resuscitation in intensive care. N Engl J Med. 2012 Nov 15;367(20):1901-11. doi: 10.1056/NEJMoa1209759. Epub 2012 Oct 17. PMID 23075127
- [Background] Navickis RJ, Haynes GR, Wilkes MM. Effect of hydroxyethyl starch on bleeding after cardiopulmonary bypass: a meta-analysis of randomized trials. J Thorac Cardiovasc Surg. 2012 Jul;144(1):223-30. doi: 10.1016/j.jtcvs.2012.04.009. Epub 2012 May 9. PMID 22578894
- [Background] Hartog CS, Reuter D, Loesche W, Hofmann M, Reinhart K. Influence of hydroxyethyl starch (HES) 130/0.4 on hemostasis as measured by viscoelastic device analysis: a systematic review. Intensive Care Med. 2011 Nov;37(11):1725-37. doi: 10.1007/s00134-011-2385-z. Epub 2011 Oct 12. PMID 21989733
- [Background] Schramko AA, Suojaranta-Ylinen RT, Kuitunen AH, Kukkonen SI, Niemi TT. Rapidly degradable hydroxyethyl starch solutions impair blood coagulation after cardiac surgery: a prospective randomized trial. Anesth Analg. 2009 Jan;108(1):30-6. doi: 10.1213/ane.0b013e31818c1282. PMID 19095827
- [Background] Akkucuk FG, Kanbak M, Ayhan B, Celebioglu B, Aypar U. The effect of HES (130/0.4) usage as the priming solution on renal function in children undergoing cardiac surgery. Ren Fail. 2013;35(2):210-5. doi: 10.3109/0886022X.2012.747139. Epub 2012 Dec 11. PMID 23228215
- [Background] Alavi SM, Ahmadi BB, Baharestani B, Babaei T. Comparison of the effects of gelatin, Ringer's solution and a modern hydroxyl ethyl starch solution after coronary artery bypass graft surgery. Cardiovasc J Afr. 2012 Sep;23(8):428-31. doi: 10.5830/CVJA-2012-026. PMID 23044498